CLINICAL TRIAL: NCT05539287
Title: Clinical Study Evaluating the Safety of Lactobacillus Probiotic in Children With Drug Resistant Epilepsy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Amira Roshdy, Assistant Lecturer of Clinical Pharmacy, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Lactobacillus in DRE.
Record Dates: First submitted 2022-09-10; First posted 2022-09-14 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2023-08

CONDITIONS: Drug Resistant Epilepsy
Keywords: Lactobacillus
MeSH Terms: conditions — Drug Resistant Epilepsy | interventions — Lacteol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Placebo Comparator): 25 patients will receive standard antiepileptic drug plus placebo capsules for 6 months.
  Interventions: Drug: Lactobacillus-Based Capsule
- Probiotic Group (Experimental): 25 patients will receive Lactobacillus species 5 billion colony forming unit (CFU) 2 capsules daily together with their standard antiepileptic drug for 6 months.
  Interventions: Drug: Lactobacillus-Based Capsule

INTERVENTIONS:
Drug: Lactobacillus-Based Capsule — 25 patients will receive Lactobacillus species 5 billion colonies forming unit (CFU) 2 capsules daily together with their standard antiepileptic drug for 6 months.
  Other Names: Lactobacillus

SUMMARY:
Animal and human studies have brought up evidence supporting Gut microbial disbalance, namely dysbiosis, as a causative factor of epilepsy, especially the refractory form. thus, probiotics might constitute a safe, low-cost, and effective supplementary therapy in patients with DRE.

The Lactobacillus population is probiotic bacteria that have a beneficial role in epilepsy. Lactobacillus can influence brain function through the modulation of GABA, as shown in rodent models. Moreover, it has been demonstrated in animal models of epilepsy and in human epileptic patients that probiotic treatment aimed at restoring gut microbiota equilibrium has beneficial effects on epileptic symptoms by increasing GABA in animals and the levels of Bifidobacteria and Lactobacillus in humans.

DETAILED DESCRIPTION:
This study will be a placebo-controlled, double-blind, and parallel 6-month duration study

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 3-18 years with intractable childhood-onset epilepsy.

  * All patients are diagnosed to have drug-resistant epilepsy (refractory epilepsy) according to the ILAE definition.
  * The subject is willing and able to comply with the study requirements

Exclusion Criteria:

* Any metabolic conditions that might increase the risks associated with trial participation or investigational product administration, such as hepatic enzyme elevation greater than twice normal and/or a GFR < 60 mL/min/1.73 m2 or electrolyte imbalance.

  * Patients who are currently using or used antibiotics therapy in the preceding month
  * Patients who are currently using or used other probiotic products in the preceding two weeks
  * Patients scheduled to undergo GIT surgery or those who underwent GIT surgery
  * Patients with a Known allergy to probiotics.
  * Patients receiving artificial enteral or intravenous nutrition

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2022-09-25 (Actual); Primary Completion 2024-08-05 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
effectivness of Lactobacillus probiotics for controlling epileptic seizures in children with drug resistant epilepsy | 6 months
  effectivness can be defined as more than 50% reduction in number of seizures.

SECONDARY OUTCOMES:
1. the change in the concentration of measured biological parameters (NLRP3, and GAD-Ab) | 6 months
  Before and 6 months after intervention, 5 ml of venous blood will be withdrawn from each participant by antecubital venipuncture between 8 am and 11 am. Blood samples will be centrifuged at 3000 rpm for 15 min to separate sera. Sera will be kept at deep freeze (-80°C) until analysis of serum concentrations of :
  * Serum NLRP3 inflammasome level.
  * Serum glutamic acid decarboxylase antibody (GAD-Ab).

CONTACTS AND LOCATIONS:
Overall Officials: tarek mostafa, professor, Study Director — Tanta University; Amira Rashdan, Rashdan, Principal Investigator — Tanta University
Locations (1):
- Amira, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: No